CLINICAL TRIAL: NCT05808400
Title: Clinical Study of the Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Exosomes in Treating Chronic Cough After COVID-19 Infection
Brief Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Exosomes in Treating Chronic Cough After COVID-19
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: REGEN-αGEEK (SHENZHEN) MEDICAL TECHNOLOGY CO., LTD. (Unknown)
Responsible Party: Principal Investigator, Jihui Du, Professor, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20230214-V04
Record Dates: First submitted 2023-04-07; First posted 2023-04-11 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Long COVID-19 Syndrome
Keywords: COVID-19; Chronic Cough
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Chronic Cough

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exosomes treatment group (Experimental): Treated with umbilical cord mesenchymal stem cell-derived extracellular vesicles (EVs) preparation (Specification: 5ml, EV concentration of 1*10^9 particles /ml)
  Interventions: Biological: MSC-derived exosomes
- Non-treatment group (No Intervention): No treatment

INTERVENTIONS:
Biological: MSC-derived exosomes — The total volume of MSC-derived exosomes is 5ml, and exosome concentration in preparation is 1*10^9 particles/ml.
  Arms: Exosomes treatment group

SUMMARY:
This clinical trial aims to evaluate the safety and effectiveness of umbilical cord mesenchymal stem cell (UCMSC)-derived extracellular vesicle nebulization inhalation therapy for the treatment of chronic cough after COVID-19 infection. The main objective is to assess whether UCMSC-derived exosome nebulization inhalation therapy alleviates chronic cough after COVID-19.

Participants will be asked to complete a questionnaire to help researchers evaluate their cough severity and to record their scores before nebulization inhalation of UCMSC-derived exosomes. Participants will receive either continuous nebulized inhalation of UCMSC-derived exosomes for 5 days, twice daily, or no treatment. Researchers will compare the experimental and control groups to evaluate the safety and efficacy of UCMSC-derived exosomes for the treatment of chronic cough after COVID-19 infection.

DETAILED DESCRIPTION:
1. Background 1.1 Post-COVID-19 Syndrome, also known as Long Covid, is still causing great trouble to the public despite China having successfully passed the first wave of infection caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) for over three years, which has resulted in over 5 million deaths globally.

   Long Covid is a multiple-system disease that includes a variety of severe symptoms that persist after infection with COVID-19, such as (1) heart-related symptoms: chest pain, palpitations; (2) respiratory symptoms: cough, shortness of breath, loss of taste or smell; (3) pancreatic symptoms: diabetes, pancreatic injury; (4) immune system: autoimmunity, mast cell activation syndrome MCAS; (5) neurological symptoms: cognitive impairment (brain fog), fatigue, sleep disorders, memory loss, tinnitus; (6) vascular symptoms: fatigue, coagulation disorders, deep vein thrombosis, endothelial dysfunction, microvascular disease, stroke; (7) reproductive symptoms: erectile dysfunction, menstrual disorders, etc., which severely affect the patient's daily life. Long Covid can occur in people of all ages, and the likelihood of developing it is closely related to the severity of acute COVID-19 infection. The main high-risk factors that can trigger Long Covid include (1) type II diabetes, (2) high viral load during COVID-19 infection, (3) previous infection with EB virus, and (4) excessive specific autoantibodies. Treatment strategies for COVID-19 mainly involve using antiviral drugs to block the replication cycle of the virus and various methods to suppress host inflammation to improve symptoms. Currently, the conventional immunotherapy methods used in clinics mainly involve the use of hormones, monoclonal antibody drugs, etc., but they are mainly targeted at more severe inflammatory reactions and suffer from low bioavailability, high cost, and significant side effects, making them unsuitable for the treatment of long COVID. Therefore, developing new immune-regulating methods with low side effects and costs would be significant for the treatment of long COVID.

   1.2 Mesenchymal stem cells (MSCs) MSCs have been shown to have comprehensive and powerful immune-regulatory and regenerative functions. MSCs can counteract cell death related to the pathogenesis of chronic obstructive pulmonary disease (COPD), idiopathic pulmonary fibrosis, asthma, ARDS, and pulmonary hypertension, and promote cell regeneration. Exosomes are one of the key paracrine effectors secreted by MSCs, and they are considered powerful candidates for alternative treatment of various diseases because their biological material is like that of progenitor cells, and they have the ability to maintain healing properties. Under physiological and pathological conditions, exosomes play a critical role in intercellular communication by transporting various biomolecules (such as miRNA and proteins) into target cells.

   1.3 the mechanism of MSC-derived exosomes MSC-derived exosomes inherit immunosuppressive properties from their source cells. MSC-EVs may use multiple mechanisms to balance the function of the immune system. One key mechanism is reprogramming and changing the phenotype of various immune cells.

   In multiple models, MSC-exosomes have therapeutic properties similar to MSCs and are easier to prepare, store, and transport to the bedside, while avoiding some limitations of cell therapy, such as the risk of pulmonary embolism and tumor formation. Exosomes secreted by MSCs can regulate immunity through an interaction with immune cells and inhibit inflammatory reactions through cytokines. Numerous studies have shown that exosomes secreted by MSCs can be used to treat immunodeficiency, inflammation, ARDS, and other lung diseases, so exosomes secreted by MSCs may also be effective in treating COVID-19 infections and pneumonia. The conventional method of stem cell therapy is an intravenous injection, and exosomes are one of the main active components secreted by stem cells with a size of 30-150 nm. After nebulization, exosomes can directly reach the bronchioles and alveoli, which is conducive to maximizing drug absorption.

   1.4 Clinical cases of MSC-derived exosomes therapy China has also actively launched relevant clinical studies. A clinical study at Wuxi Fifth People's Hospital in Jiangsu Province confirmed that nebulized umbilical cord mesenchymal stem cell-derived exosomes are safe and feasible for treating COVID-19 pneumonia. Researchers at Ruijin Hospital and Jin Yin-tan Hospital jointly conducted nebulized exosome therapy for COVID-19 using exosomes derived from human allogeneic adipose mesenchymal stem cells (HAMSCs-Exos). Recently, the inhaled anti-COVID-19 drug Exo-CD24, a combination of exosomes and CD24 protein, has shown promising results in phase I clinical trial led by Israeli medical center expert Nadir Arber. Out of 30 critically ill volunteers in the trial, 29 were cured after five days of treatment. Although Exo-CD24 has yet to pass phase III testing, it has already demonstrated enormous potential for the future. The US FDA has approved Direct Biologics to start a phase I/II trial to evaluate ExoFlo™ for treating COVID-19. This marks the first time that extracellular vesicles (EVS) have been approved by the US FDA for treating the disease.
2. Research Purpose The aim of this study is to evaluate the safety and effectiveness of umbilical cord mesenchymal stem cell exosome nebulization inhalation for treating chronic cough in patients after COVID-19 infection through a non-randomized controlled clinical trial.
3. Study Design The study design is a prospective, non-randomized, concurrent controlled trial. Based on the routine treatment regimen for COVID-19 infection according to clinical guidelines, umbilical cord mesenchymal stem cell exosome nebulization inhalation will be used in the experimental group to treat chronic cough in patients after COVID-19 infection. The experimental group (n=40) and control group (n=40) will be compared with patients who did not receive exosome nebulization inhalation therapy during the same period. The safety and effectiveness of umbilical cord mesenchymal stem cell exosome nebulization inhalation for treating chronic cough in patients after COVID-19 infection will be evaluated through cough severity score surveys, symptom improvement time, and adverse event occurrence.

3.1 Study Population A total of 80 participants will be enrolled in the study, with a ratio of 1:1 for the experimental group (n=40) and the control group (n=40). The study population will consist of COVID-19-infected patients who meet the selection criteria and are treated in the COVID-19 rehabilitation outpatient clinic at the Shenzhen Hospital of Southern Medical University.

3.2 Grouping (1) Experimental group: Nebulization inhalation of umbilical cord mesenchymal stem cell exosome preparation; specification: 5ml, exosome concentration in preparation is 1*10^9 particles/ml.

(2) Control group: Patients during the same period who did not receive treatment with stem cell exosomes.

ELIGIBILITY:
Inclusion Criteria:

* Trial participants voluntarily participate in this study and sign an informed consent form.
* At the time of signing the informed consent form, the age of the subject should be ≥18 or ≤80 years old, with no gender restrictions.
* The subject has been diagnosed with COVID-19 (confirmed by positive nucleic acid or antigen test) and has symptoms that have lasted for more than 4 weeks.
* Negative nucleic acid or antigen test at the time of screening.
* The subject has had continuous or intermittent coughing, or loss of taste/smell for ≥4 weeks, which did not occur before the onset of COVID-19 infection.
* No prior treatment with umbilical cord mesenchymal stem cell-derived extracellular vesicles.
* The patient fully understands the purpose and requirements of this clinical study and is willing to complete all trial procedures according to the study requirements.

Exclusion Criteria:

* Age ≤18 or ≥80 years old.
* Acute COVID-19 patients.
* Suspected or confirmed to have severe, active bacterial, fungal, or other infections that may pose a risk when intervention measures are taken, as determined by the researcher.
* Patients with a history of diagnosed bronchial asthma, cough variant asthma, or chronic cough; patients with other pulmonary diseases such as chronic obstructive pulmonary disease, bronchiectasis, tuberculosis, lung cancer, etc.
* Any of the following during the screening period: 1) ALT or AST > 3 times the upper limit of normal; 2) eGFR <60 mL/min.
* Patients with a history of severe allergies.
* Patients with uncontrolled severe cardiovascular, cerebrovascular, liver, kidney, endocrine, blood system diseases, and mental illness.
* Patients with active immunosuppression, immunodeficiency, and use of immunosuppressive drugs.
* Pregnant and lactating women.
* Other factors that the researcher deems unsuitable for participation in the study based on clinical considerations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Cough Evaluation Test | 6-14days
  This score is to evaluate the relief of cough symptoms. Higher scores mean worse outcome. Minimum score is 5, maximum score is 25.

SECONDARY OUTCOMES:
Improvement or relief time of symptoms | 6th, 15th, 28th day
  This indicator is to evaluate how many days it takes to alleviate cough

OTHER OUTCOMES:
Pulmonary function tests or lung CT scans | 14th day
  This indicator is to evaluate lung function

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Du, PhD, Principal Investigator — Huazhong University of Science and Technology Union Shenzhen Hospital
Locations (1):
- Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Shennawy L, Hoffmann AD, Dashzeveg NK, McAndrews KM, Mehl PJ, Cornish D, Yu Z, Tokars VL, Nicolaescu V, Tomatsidou A, Mao C, Felicelli CJ, Tsai CF, Ostiguin C, Jia Y, Li L, Furlong K, Wysocki J, Luo X, Ruivo CF, Batlle D, Hope TJ, Shen Y, Chae YK, Zhang H, LeBleu VS, Shi T, Swaminathan S, Luo Y, Missiakas D, Randall GC, Demonbreun AR, Ison MG, Kalluri R, Fang D, Liu H. Circulating ACE2-expressing extracellular vesicles block broad strains of SARS-CoV-2. Nat Commun. 2022 Jan 20;13(1):405. doi: 10.1038/s41467-021-27893-2. PMID 35058437
- [Background] Davis HE, McCorkell L, Vogel JM, Topol EJ. Long COVID: major findings, mechanisms and recommendations. Nat Rev Microbiol. 2023 Mar;21(3):133-146. doi: 10.1038/s41579-022-00846-2. Epub 2023 Jan 13. PMID 36639608
- [Background] Davido B, Seang S, Tubiana R, de Truchis P. Post-COVID-19 chronic symptoms: a postinfectious entity? Clin Microbiol Infect. 2020 Nov;26(11):1448-1449. doi: 10.1016/j.cmi.2020.07.028. Epub 2020 Jul 23. No abstract available. PMID 32712242
- [Background] Su Y, Yuan D, Chen DG, Ng RH, Wang K, Choi J, Li S, Hong S, Zhang R, Xie J, Kornilov SA, Scherler K, Pavlovitch-Bedzyk AJ, Dong S, Lausted C, Lee I, Fallen S, Dai CL, Baloni P, Smith B, Duvvuri VR, Anderson KG, Li J, Yang F, Duncombe CJ, McCulloch DJ, Rostomily C, Troisch P, Zhou J, Mackay S, DeGottardi Q, May DH, Taniguchi R, Gittelman RM, Klinger M, Snyder TM, Roper R, Wojciechowska G, Murray K, Edmark R, Evans S, Jones L, Zhou Y, Rowen L, Liu R, Chour W, Algren HA, Berrington WR, Wallick JA, Cochran RA, Micikas ME; ISB-Swedish COVID-19 Biobanking Unit; Wrin T, Petropoulos CJ, Cole HR, Fischer TD, Wei W, Hoon DSB, Price ND, Subramanian N, Hill JA, Hadlock J, Magis AT, Ribas A, Lanier LL, Boyd SD, Bluestone JA, Chu H, Hood L, Gottardo R, Greenberg PD, Davis MM, Goldman JD, Heath JR. Multiple early factors anticipate post-acute COVID-19 sequelae. Cell. 2022 Mar 3;185(5):881-895.e20. doi: 10.1016/j.cell.2022.01.014. Epub 2022 Jan 25. PMID 35216672
- [Background] Carrade Holt DD, Wood JA, Granick JL, Walker NJ, Clark KC, Borjesson DL. Equine mesenchymal stem cells inhibit T cell proliferation through different mechanisms depending on tissue source. Stem Cells Dev. 2014 Jun 1;23(11):1258-65. doi: 10.1089/scd.2013.0537. Epub 2014 Mar 4. PMID 24438346
- [Background] Sauler M, Bazan IS, Lee PJ. Cell Death in the Lung: The Apoptosis-Necroptosis Axis. Annu Rev Physiol. 2019 Feb 10;81:375-402. doi: 10.1146/annurev-physiol-020518-114320. Epub 2018 Nov 28. PMID 30485762
- [Background] Naji A, Suganuma N, Espagnolle N, Yagyu KI, Baba N, Sensebe L, Deschaseaux F. Rationale for Determining the Functional Potency of Mesenchymal Stem Cells in Preventing Regulated Cell Death for Therapeutic Use. Stem Cells Transl Med. 2017 Mar;6(3):713-719. doi: 10.5966/sctm.2016-0289. Epub 2016 Oct 11. PMID 28297565
- [Background] Janockova J, Slovinska L, Harvanova D, Spakova T, Rosocha J. New therapeutic approaches of mesenchymal stem cells-derived exosomes. J Biomed Sci. 2021 May 25;28(1):39. doi: 10.1186/s12929-021-00736-4. PMID 34030679
- [Background] Joo HS, Suh JH, Lee HJ, Bang ES, Lee JM. Current Knowledge and Future Perspectives on Mesenchymal Stem Cell-Derived Exosomes as a New Therapeutic Agent. Int J Mol Sci. 2020 Jan 22;21(3):727. doi: 10.3390/ijms21030727. PMID 31979113
- [Background] Modani S, Tomar D, Tangirala S, Sriram A, Mehra NK, Kumar R, Khatri DK, Singh PK. An updated review on exosomes: biosynthesis to clinical applications. J Drug Target. 2021 Nov;29(9):925-940. doi: 10.1080/1061186X.2021.1894436. Epub 2021 Mar 12. PMID 33709876
- [Background] Morrison TJ, Jackson MV, Cunningham EK, Kissenpfennig A, McAuley DF, O'Kane CM, Krasnodembskaya AD. Mesenchymal Stromal Cells Modulate Macrophages in Clinically Relevant Lung Injury Models by Extracellular Vesicle Mitochondrial Transfer. Am J Respir Crit Care Med. 2017 Nov 15;196(10):1275-1286. doi: 10.1164/rccm.201701-0170OC. PMID 28598224
- [Background] Wu P, Zhang B, Shi H, Qian H, Xu W. MSC-exosome: A novel cell-free therapy for cutaneous regeneration. Cytotherapy. 2018 Mar;20(3):291-301. doi: 10.1016/j.jcyt.2017.11.002. Epub 2018 Feb 9. PMID 29434006
- [Background] Chu M, Wang H, Bian L, Huang J, Wu D, Zhang R, Fei F, Chen Y, Xia J. Nebulization Therapy with Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes for COVID-19 Pneumonia. Stem Cell Rev Rep. 2022 Aug;18(6):2152-2163. doi: 10.1007/s12015-022-10398-w. Epub 2022 Jun 4. PMID 35665467

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT05808400/Prot_SAP_ICF_000.pdf